CLINICAL TRIAL: NCT01590550
Title: A Prospective Study of Citrate Based Dialysate in Pediatric Patients Receiving Intermittent Hemodialysis
Brief Title: Observational Study of Citrate Based Dialysis in Pediatric Patients Receiving Hemodialysis
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Rita Sheth, Assistant Professor - Pediatrics, Loma Linda University
Other Study IDs: 5120017
Record Dates: First submitted 2012-04-29; First posted 2012-05-03 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Complication of Dialysis
Keywords: Pediatric hemodialysis; Anticoagulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single arm: Single arm for all patient receiving inpatient HD
  Interventions: Procedure: Use of citrate based dialysate

INTERVENTIONS:
Procedure: Use of citrate based dialysate — Use of heparin free citrate based dialysate

SUMMARY:
Providing hemodialysis requires the use of an extracorporeal circuit which must be anticoagulated. Inadequate anticoagulation can result in the dialyzer clotting with decreased circuit blood flows, inefficient dialysis and even significant blood loss secondary to circuit clotting.Heparin has been traditional agent used to provide anticoagulation. Heparin has multiple adverse side effects that would be best avoided in acutely ill patients who are at risk for bleeding. Alternative means of providing anticoagulation include citrate based anticoagulation. Citrasate® is a heparin free anticoagulant alternative that has been FDA approved since 1999 and readily available for commercial use since 2001. Citrasate® utilizes citric acid instead of acetic acid for acidification; the presence of small amounts of citrate in the dialysate also provides the means for anticoagulation. The concentration of citrate is low (2.4meq/L) and thus has a minimal effect on serum calcium values. No calcium monitoring or infusion is indicated.

The purpose of this study is to obtain further data on the use of Citrasate® in admitted pediatric patients who receive hemodialysis as part of their therapy for acute kidney injury.

DETAILED DESCRIPTION:
All patients requiring inpatient hemodialysis will be screened for participation in the study based on inclusion and exclusion criteria as noted above. Informed consent for hemodialysis and for study participation will be obtained by the attending nephrologist prior to the start of the dialysis session. Patient specific hemodialysis orders will be placed by attending nephrology physician for each patient using a standardized hemodialysis order form. Citrasate® in standard concentration, with a standard blood flow of 600 -800 ml/min will be prescribed for all study patients, calcium and potassium contents of the dialysate will be determined by the attending pediatric nephrologist.

Monitoring: All patients will have routine monitoring as indicated for clinical care during each dialysis session.

Data Collection:Each treatment will be documented on a standardized hemodialysis run sheet. Data collection will be performed by any one of the researchers using a data collection sheet to ensure uniformity of data collection methods. Data to be collected includes patient demographics, admitting diagnosis, underlying renal disease, the presence of acute kidney injury versus chronic kidney disease, contraindications to heparin use and the presence of any bleeding diathesis. Dialysis specific data to be collected will include the site and type of dialysis access, dialysis prescription parameters and treatment duration. Lab data to be collected will include pre, post and intradialytic ionized calcium values, ACT values and pH and bicarbonate values. Data on the number of saline boluses required to maintain circuit patency, percent of prescribed blood flow achieved as well as any use of heparin will be collected.

Data Analysis will include

* T-test for comparison of changes in ionized calcium values, blood pH and bicarbonate values
* Percentage of patients with inadequate coagulation on citrate (ie. patients with grade III-IV streaking or required changing to heparin based dialysate)
* Percent of patients with any adverse events not accounted for during an routine dialysis session
* Cost analysis for the difference in costs using Citrasate® compared to a standard heparin based dialysis treatment

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients between the ages of 0-21 years in the inpatient setting requiring hemodialysis for renal replacement therapy. These will include both patients with chronic renal failure and acute kidney injury, or any patient requiring dialysis as determined by an attending nephrologist.

Exclusion Criteria:

* Symptomatic hypocalcemia that is refractory to treatment 24 hours prior to the start of each dialysis session
* Known liver disorder/acute liver failure with an inability to metabolize citrate.

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Admitted pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita D Sheth, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Children's Hospital, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No
Mean data will be presented

REFERENCES:
- [Background] Hanevold C, Lu S, Yonekawa K. Utility of citrate dialysate in management of acute kidney injury in children. Hemodial Int. 2010 Oct;14 Suppl 1:S2-6. doi: 10.1111/j.1542-4758.2010.00483.x. PMID 21040414
- [Background] Davenport A. Anticoagulation options for pediatric hemodialysis. Hemodial Int. 2003 Apr 1;7(2):168-76. doi: 10.1046/j.1492-7535.2003.00022.x. PMID 19379358
- [Background] Cheng YL, Yu AW, Tsang KY, Shah DH, Kjellstrand CM, Wong SM, Lau WY, Hau LM, Ing TS. Anticoagulation during haemodialysis using a citrate-enriched dialysate: a feasibility study. Nephrol Dial Transplant. 2011 Feb;26(2):641-6. doi: 10.1093/ndt/gfq396. Epub 2010 Jul 8. PMID 20615906
- [Background] Gabutti L, Lucchini B, Marone C, Alberio L, Burnier M. Citrate- vs. acetate-based dialysate in bicarbonate haemodialysis: consequences on haemodynamics, coagulation, acid-base status, and electrolytes. BMC Nephrol. 2009 Mar 5;10:7. doi: 10.1186/1471-2369-10-7. PMID 19265544

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric patients receiving hemodialysis (HD) at a single institution during the specified study period
Groups:
- Observational: All patients receiving acute HD during the study period
Period: Overall Study
Arm/Group | Observational
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Observational
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Dialyzer Clotting Rate
Description: Dialyzer clotting rate will be assessed as the percent of hemodialysis treatments that developed a clot in the dialyzer from the time that the patient is enrolled in the study until the time hemodialysis treatments with Citrasate® are discontinued.
Time Frame: Followed until HD with Citrate dialysate is discontinued, average 3 weeks
Population: 18 patients and 119 HD treatments
Measure: Number; unit: percentage of total treatments
Groups:
- Observational: All patients receiving acute HD during the study period 6/118 (5%) treatments with circuit or catheter clotting
Arm/Group | Observational
Number analyzed (Participants) | 18
percentage of total treatments | 6

2. Secondary Outcome: Saline Flush Rate
Description: Saline flush rate will be assesed as the percentage of hemodialysis treatments that require one or more saline flushes to maintain circuit patency from the time that the patient is enrolled in the study until the time hemodialysis treatments with Citrasate® are discontinued based on clinical indications, upto a maximum period of 6 months
Time Frame: Patients will be followed until HD Citrate dialysate is discontinued, average 3 weeks
Measure: Number; unit: percentage of hemodialysis treatments
Arm/Group | Observational
Number analyzed (Participants) | 18
percentage of hemodialysis treatments | 0

3. Secondary Outcome: Heparin Use Rate
Description: The heparin use rate will be assessed as the percentage of hemodialysis treatments that required additional use of heparin to maintain circuit patency. This will be assessed from the time that the patient is enrolled in the study until the time hemodialysis treatments with Citrasate® are discontinued based on clinical indications, upto a maximum period of 6 months
Time Frame: Patients will be followed until inpatient hemodialysis sessions with Citrasate® are discontinued
Measure: Number; unit: percentage of hemodialysis treatments
Arm/Group | Observational
Number analyzed (Participants) | 18
percentage of hemodialysis treatments | 0

ADVERSE EVENTS:
Arm/Group | Observational
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 3/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational (N=18)
Clotting of circuit (General disorders) | 3 (6) — Clotting of extracorporeal circuit

LIMITATIONS AND CAVEATS:
No control group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes